CLINICAL TRIAL: NCT05463575
Title: Metabolic Effects of Ketohexokinase Inhibition on Individuals With Non-alcoholic Fatty Liver Disease
Brief Title: Ketohexokinase Inhibition in NAFLD
Acronym: KHKi
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NL80131.068.22 / METC 22-006
Record Dates: First submitted 2022-07-01; First posted 2022-07-19 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: NAFLD
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PF-06835919 (Experimental): KHKi
  Interventions: Drug: Ketohexokinase inhibition
- Placebo (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Ketohexokinase inhibition — participants will be asked to take 300 mg of the KHKi in tablet form daily for 6 weeks in either period 1 or 2.
  Arms: PF-06835919
Other: Placebo — participants will be asked to take 300 mg of the placebo in tablet form daily for 6 weeks in either period 1 or period 2.
  Arms: Placebo

SUMMARY:
Fructose is a big contributor to the development of non-alcoholic fatty liver disease (NAFLD). Inhibiting ketohexokinase (KHK), the enzyme catalyzing the first committed step in fructose metabolism, is thought to reduced intrahepatic lipid (IHL) content. Pharmacological inhibition of KHK resulted in a decrease in IHL content in NAFLD patients, but additional health effects are still unknown. In this study the investigators aim to look at additional health effects following KHK inhibition (KHKi).

DETAILED DESCRIPTION:
Rationale: NAFLD is a highly prevalent (~30%) disease that is histologically characterized by simple steatosis, steatohepatitis and/or fibrosis in the absence of alcohol abuse. Liver fibrosis can progress to cirrhosis, which is a risk factor for endstage liver disease and hepatocellular carcinoma. Of interest, recent studies have shown that NAFLD is also a risk factor for systemic diseases, such as type 2 diabetes, which is probably mediated by hepatic insulin resistance. Previous research showed that inhibition of KHK, the first step in fructose metabolism, reduces IHL content in individuals with NAFLD. KHK is predominantly expressed in the gut, kidney, and liver where it facilitates the phosphorylation of fructose to fructose-1P, and thereby entrapment and subsequent metabolism within the cell. KHKi in the liver, therefore, impairs entrapment of ingested fructose and, consequently, conversion into fat which might lead to improvements in hepatic insulin sensitivity. However, studies investigating the effect of KHKi on hepatic insulin sensitivity are lacking. Objective: The primary objective of this study is to assess the effect of KHKi on hepatic insulin sensitivity in overweight/obese individuals with non-alcoholic fatty liver disease. The secondary objective includes the assessment of KHKi on fat distribution, adipose tissue insulin sensitivity, and fat oxidation in overweight/obese individuals with non-alcoholic fatty liver disease.

Explorative objectives are the assessment of in vivo KHK activity, gut microbiota composition and alternative metabolic pathways upon KHK inhibition. Study design: The present study is a randomized, double-blinded, placebo-controlled cross over trial (RCT).

Study population: 14 overweight/obese (BMI: 27-35 kg/m2

), male and (postmenopausal) female participants, aged 45 - 70 years with non-alcoholic fatty liver disease (IHL ≥ 5.56%) will participate in this study. From experience with similar studies, the investigators estimate a drop-out rate of 20% and a screening failure of 50% (due to the strict inclusion criteria), resulting in maximally 17 subjects that have to be included and 36 subjects that have to be screened (maximally).

Intervention (if applicable): Participants receive once daily (in the morning) 300 mg in tablet form.

of the KHK inhibitor PF-06835919 or a placebo for 42 days. Main study parameters/endpoints: The primary study endpoint is hepatic insulin sensitivity measured during a hyperinsulinemic-euglycemic clamp. Secondary outcome parameters are fat distribution, adipose tissue insulin sensitivity and fat oxidation. Explorative objectives are in vivo KHK activity, gut microbiota composition, and alternative metabolic pathways.

Nature and extent of the burden and risks associated with participation, benefit, and group relatedness: PF-06835919 is well-tolerated and has not been associated with major side-effects. The main burden of this study is the large time investment. During the intervention

periods, subjects will receive once daily (in the morning) 300 mg of the KHK inhibitor During the last three days of each intervention period, participants visit to the research facility for a 2-day stay (with overnight stay) for the test measurements (total time investment per intervention period is 34 hours). Moreover, the test days comprise several non-invasive and invasive measurements. The used techniques are safe, but the muscle biopsies can cause some discomfort and may result in a local bruise or hematoma. Likewise, blood sampling can cause a local hematoma. The risk of infection and/or prolonged bleeding is very low due to state-of-the-art techniques and sterility measures. During the hyperinsulinemic-euglycemic clamp, a very small risk of hypoglycaemia exists. In summary, we will draw approximately 184ml blood during the entire study period. Measurements performed during the time course of the study can potentially lead to unexpected medical findings. Subjects will be informed about such a finding and possible advised to contact a doctor about this. If a subject does not want to be informed about incidental findings, participation in this study is not possible.

ELIGIBILITY:
Inclusion Criteria:

* Participants are able to provide signed and dated written informed consent prior to any study specific procedures
* Men and (postmenopausal) woman
* Aged ≥ 45 and ≤ 70 years
* Body mass index (BMI) 27 - 35 kg/m2
* Hepatic steatosis (i.e. IHL ≥ 5.56%)
* Stable dietary habits (no weight loss or gain > 3 kg in the past 3 months)

Exclusion Criteria:

* Type 2 diabetes
* Patients with congestive heart failure and and/or severe renal and or liver insufficiency
* Uncontrolled hypertension
* Any contra-indication for MRI scanning
* Alcohol consumption of >3 servings per day for man and >2 servings per day for woman
* Smoking
* Unstable body weight (weight gain or loss > 3kg in the last 3 months)
* Engagement in structured exercise activities > 2 hours a week
* Previous enrolment in a clinical study with an investigational product during the last 3 months or as judged by the investigator which would possibly hamper our study results
* Use of drugs that inhibit organic anion transporting polypeptide (OATP) transporters (e.g. rifampicin, gemfibrozil, cyclosporine, erythromycin and clarithromycin)
* Subjects who do not want to be informed about unexpected medical findings

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-11-24 (Actual); Study Completion 2023-11-24 (Actual)

PRIMARY OUTCOMES:
Hepatic insulin sensitivity | 42 days
  insulin-mediated suppression of endogenous glucose production (EGP) in µmol/kg/min measured during the 2- step hyperinsulinemic-euglycemic clamp

SECONDARY OUTCOMES:
Intrahepatic lipid content | 41 days
  1H-MRS in percent
Liver lipid content composition | 41 days
  1H-MRS in percent
Subcutaneous adipose tissue | 41 days
  MRI in cm^3
Visceral adipose tissue | 41 days
  MRI in cm^3
Insulin-mediated suppression of free fatty acids | 42 days
  Plasma in mmol/L
Inflammatory markers like adiponectin, interleukin-6, hsCRP, TNF-α | 42 days
  in blood serum in µg/mL
Resting energy expenditure (REE) | 42 days
  kcal/kg/min
Sleeping metabolic rate | 42 days
  kcal/kg/min
Body composition | 42 days
  fat mass (kg and percent)
Body composition | 42 days
  fat-free mass (kg and percent)

OTHER OUTCOMES:
Liver phosphomonoester levels | 41 days
  31P-MRS in mg/kg bw after an oral fructose load as a measure of KHK activity
Peripheral insulin sensitivity | 42 days
  Rd during the clamp in µmol/kg/min
Metabolic flexibility | 42 days
  delta REE between basal and insulin stimulated state
Intramyocellular lipid content | 42 days
  measured in muscle biopsies in arbitrary units
Fecal short-chain fatty acids including acetate, propionate, and butyrate | 41 days
  concentration in fecal samples in μmol/g

CONTACTS AND LOCATIONS:
Locations (1):
- Maastricht University Medical centre, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: No
Data can be obtained with the PI on request